CLINICAL TRIAL: NCT02300740
Title: Pharmacokinetic Analysis of Nicotinamide Riboside
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Britt Christensen, Cand.Scient, PhD, Post doc, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 45141
Record Dates: First submitted 2014-11-20; First posted 2014-11-25 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Participants
MeSH Terms: interventions — nicotinamide-beta-riboside

ARMS (2):
- low dose (Experimental): 500 mg nicotinamide riboside oral
  Interventions: Dietary Supplement: Nicotinamide riboside
- high dose (Experimental): 1000 mg nicotinamide riboside oral
  Interventions: Dietary Supplement: Nicotinamide riboside

INTERVENTIONS:
Dietary Supplement: Nicotinamide riboside — NIAGEN, ChromaDex

SUMMARY:
Nicotinamide riboside is a newly discovered vitamin B3. The pharmacokinetics in humans is so far not analyzed.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-25, healthy, male,

Exclusion Criteria:

* liver or kidney diseases, other diseases

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Serum nicotinamide riboside | 8 hours, blood samples every 15 min

SECONDARY OUTCOMES:
serum concentrations of metabolites of nicotinamide riboside | 8 hour, blood samples every 15 min
area under the curve for serum nicotinamide riboside | 8 hours, blood samples every 15 min
calculation of halftime of serum nicotinamide riboside | 8 hours, blood samples every 15 min
calculation of C-max of serum nicotinamide riboside | 8 hours, blood samples every 15 min
calculation of t-max of serum nicotinamide riboside | 8 hours, blood samples every 15 min

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Research Laboratories, Aarhus University Hospital, Aarhus, Denmark